CLINICAL TRIAL: NCT02962999
Title: Effect Of Ketamine Infusion On Oxygenation And Ventilation Mechanics In Patients With Chronic Obstructive Pulmonary Disease Applied One Lung Ventilation
Brief Title: Effect Of Ketamine Infusion In Patients With COPD Applied One Lung Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Feride Karacaer, Specialist doctor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KCOPD1
Record Dates: First submitted 2016-10-31; First posted 2016-11-15 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease Mild; Chronic Obstructive Pulmonary Disease Moderate; Chronic Obstructive Pulmonary Disease Severe; Lungcancer; Anesthesia
Keywords: Ketamine; One lung ventilation; Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): After induction, patients will be received 1 mg/kg ketamine bolus, then will be administered 0,5 mg/kg/hour ketamine infusion intraoperatively. Anesthesia will be maintained with %4-6 desflurane and 0,25-0,5 microgram/dk/min remifentanil.
  Interventions: Drug: Ketamine
- Saline (Placebo Comparator): After induction, patients will be received saline bolus, then will be administered saline infusion intraoperatively. Anesthesia will be maintained with %4-6 desflurane and 0,25-0,5 microgram/dk/min remifentanil.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — After induction, patients will be received 1 mg/kg ketamine bolus, then administered 0,5 mg/kg/hour ketamine infusion intraoperatively.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Saline — After induction, patients will be received saline bolus, then will be administered saline infusion intraoperatively.
  Other Names: %0,9 NaCl
  Arms: Saline

SUMMARY:
Chronic obstructive pulmonary disease (COPD) patients often undergo thoracic surgery due to lung cancer and emphysematous changes. One lung ventilation (OLV) used in thoracic surgery aggravates hypoxia and hypercapnia increasing intrapulmonary shunt and dead space.Ketamine provide bronchodilation by inhibiting the reuptake of catecholamines in the circulation. It also serves relaxation of bronchial smooth muscle. Our aim in this study, effects of ketamine on arterial oxygenation, the shunt fraction and the lung mechanics in patients with COPD who administered OLV because of thoracic surgery. Thirty patients with COPD who undergo thoracotomy for lung lobectomy will be included in this study. Patients will be randomly divided to a control group (%0,9 saline- CG) or a keta (ketamine- KG) group. KG will be administered 1 mg/kg ketamine bolus, then 0,5 mg/kg/hour ketamine infusion after the induction, CG will be administered sline bolus, then saline infusion. Peak airway pressure (Ppeak), plato airway pressure (Pplato), static compliance, shunt fraction, PaO2/FiO2 and arteriel blood gas values (Pa02, PaC02) will be recorded before initiation of OLV and 30 minutes intervals after initiation of OLV.To evaluate the postoperative pulmonary complications, Pa02, PaC02 in blood gas and Pa02/Fi02 values will be recorded 20 minute after arrival at postoperative care unit. Patients will be evaluated for pneumonia, atelectasis and acute lung injury at postoperative 72 h and findings will be recorded. 30 day mortality will be recorded.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a risk factor for cardiopulmonary morbidity and mortality after thoracic surgery. The elastic recoil reduction and structural changes in the small airways and alveoli cause pulmonary air trapping and hyperinflation in patients with COPD. Chronic alveolar hypoxia results structural changes in the pulmonary arteriol such as medial hypertrophy and muscularization. Ventilation-perfusion mismatch and from the right to left shunt cause hypoxia in patients with COPD. COPD patients often undergo thoracic surgery due to lung cancer and emphysematous changes. One lung ventilation (OLV) used in thoracic surgery aggravates hypoxia and hypercapnia increasing intrpulmonary shunt and dead space. Positive end expirium pressure (PEEP) and alveolary recruitment are not applicable to treat hypoxia because of development of high intrinsic PEEP. Ketamine is an intravenous general anesthetic agent widely used for many years and has sympathomimetic bronchodilator features on the airway. Ketamine provide bronchodilation by inhibiting the reuptake of catecholamines in the circulation. It also serves relaxation of bronchial smooth muscle. Our aim in this study, effects of ketamine on arterial oxygenation, the shunt fraction and the lung mechanics in patients with COPD who administered OLV because of thoracic surgery. This prospective, randomized, double blinded, controlled study will be conducted following Cukurova University Faculty of Medicine Ethics Committee approval and written informed patient consent. Thirty patients who undergo thoracotomy for lung lobectomy will be included in this study.Patients will be monitored for electrocardiography (ECG), oxygen saturation (Sa02) and non-invasive blood pressure and applied thoracal (T 5-8) epidural catheter which will be used postoperative analgesia. After the induction of anesthesia, patients will be intubated with double lumen tube (DLT). The position of the DLT will be confirmed with fiberoptic bronchoscope. Anesthesia will be maintained with %4-6 desflurane and 0,25-0,5 microgram/dk/min remifentanil. Desflurane will be titrated to maintain a bispectral index of 40 to 60.Patients will be randomly divided to a control group (%0,9 saline- CG) or a keta (ketamine- KG) group. KG will be received 1 mg/kg ketamine bolus, then 0,5 mg/kg/hour ketamine infusion will be administered until the end of operation, CG will be received bolus saline, then saline infusion will be administered until the end of operation . Patients will be ventilated with volume controlled ventilation (VCV), tidal volume (TV) 8 mlt/kg and rate of inspirium:expirium (I:E)=1:2,5 during two lung ventilation. During OLV, the lungs were ventilated with VCV, TV 5 mlt/kg, I:E=1:2,5, PEEP= 5cmH20. The fraction of inspired oxygen (Fi02) will initially set at 0,6. In cases of desaturation to Sa02 less than 95%, Fi02 will be increased by 0,2 up to 1,0. Peak airway pressure (Ppeak), plato airway pressure (Pplato), static compliance, shunt fraction and arteriel blood gas values (Pa02, PaC02) will be recorded before initiation of OLV and 30 minutes intervals after initiation of OLV. To evaluate the postoperative pulmonary complications, Pa02, PaC02 in blood gas and Pa02/Fi02 values will be recorded 20 minute after and 1 hour after arrival at postoperative care unit. If the patient shows signs of dyspnea and Pa02/Fi02<300, the patient will be admitted intensive care unit. Patients will be evaluated for pneumonia, atelectasis and acute lung injury at postoperative 72 h and findings will be recorded. 30 day mortality will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 40 years
* American Society of Anesthesiologists' physical status 2-3
* Diagnosis of COPD
* Forced expiratory volume in 1 second (FEV1) ≥ %50 in a preoperative pulmonary function test.

Exclusion Criteria:

* Heart failure
* Severe functional liver or kidney disease
* Pregnancy,
* Obesity (BMI≥30)
* Respiratory failure (Pa02< 55 mmHg, PaC02> 55 mmHg)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change of Peak airway pressure (mmHg) | From the start of OLV to end of OLV intraoperatively (before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV)
  Peak airway pressure (Ppeak-mmHg) will be recorded before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV. Change from initiation of Ppeak at 120 minute will be evaluated.

SECONDARY OUTCOMES:
Change of arteriel P02 | From the start of OLV to postoperative 1 hour.(before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV. Pa02 in blood gas values will be recorded 20 minute after arrival at postoperative care unit.
  arteriel blood gas value (Pa02-mmHg) will be recorded before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV and postoperative 1 hour. Pa02 in blood gas values will be recorded 20 minute after and 1 hour after arrival at postoperative care unit.
Change of Shunt fraction | From the start of OLV to end of OLV intraoperatively (before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV)
  Shunt fraction will be calculated with; Qs/Qt= (5,8xRI)+6,7 RI= Respiratory index RI= (PA02-Pa02)/ Pa02 PA02= Alveolar 02 pressure PA02= ([PB-PH20]x Fi02)- PaC02 PB= Atmosphere pressure= 760 mmHg PH20= Water vapor pressure= 47 mmHg shunt fraction will be recorded before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation OLV
Change of Plato airway pressure (mmHg) | From the start of OLV to end of OLV intraoperatively (before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV)
  Plato airway pressure (Pplato-mmHg) will be recorded before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV. Change from initiation of Ppeak at 120 minute will be evaluated.
Change of arteriel PC02 | From the start of OLV to postoperative 1 hour.(before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV. PaC02 in blood gas values will be recorded 20 minute after arrival at postoperative care unit.)
  arteriel blood gas value (PaC02-mmHg) will be recorded before initiation of OLV and 30 minutes intervals up to 120 minutes after initiation of OLV and postoperative 1 hour. PaC02 in blood gas values will be recorded 20 minute after and 1 hour after arrival at postoperative care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Feride Karacaer, Specialist, Study Director — Cukurova University
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University, Adana
  - Cukurova University Faculty of Medicine Research Hospital, Adana

REFERENCES:
- [Background] Weinreich AI, Silvay G, Lumb PD. Continuous ketamine infusion for one-lung anaesthesia. Can Anaesth Soc J. 1980 Sep;27(5):485-90. doi: 10.1007/BF03007049. PMID 7448609
- [Background] Rees DI, Gaines GY 3rd. One-lung anesthesia--a comparison of pulmonary gas exchange during anesthesia with ketamine or enflurane. Anesth Analg. 1984 May;63(5):521-5. PMID 6711845
- [Background] Lee SH, Kim N, Lee CY, Ban MG, Oh YJ. Effects of dexmedetomidine on oxygenation and lung mechanics in patients with moderate chronic obstructive pulmonary disease undergoing lung cancer surgery: A randomised double-blinded trial. Eur J Anaesthesiol. 2016 Apr;33(4):275-82. doi: 10.1097/EJA.0000000000000405. PMID 26716866